CLINICAL TRIAL: NCT01117025
Title: The Role of Renal Denervation in Improving Outcomes of Catheter Ablation in Patients With Refractory Symptomatic Atrial Fibrillation and Resistant Hypertension
Brief Title: Combined Treatment of Resistant Hypertension and Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDAFA-029; RU MC 001 (Other: State Research Institute of Circulation Pathology)
Record Dates: First submitted 2010-04-30; First posted 2010-05-05 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Hypertension, Resistant to Conventional Therapy; Atrial Fibrillation
Keywords: Resistant hypertension; Atrial Fibrillation; Percutaneous renal denervation
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Circumferential PVI (Active Comparator)
  Interventions: Procedure: Circumferential PV isolation
- Circumferential PVI+renal denervation (Active Comparator)
  Interventions: Procedure: Circumferential PVI+renal denervation

INTERVENTIONS:
Procedure: Circumferential PV isolation — The left atrium (LA) and pulmonary veins (PVs) are explored through a transeptal approach. Real-time 3D LA maps are reconstructed by using a nonfluoroscopic navigation system. The ipsilateral left and right PVs are encircled in one lesion line by circumferential PV isolation. Radiofrequency energy is delivered at 43°C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and is reduced to 43°C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation speed of 17 mL/min. Each lesion is ablated continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 s. The endpoint of circumferential PV isolation is PV isolation. Additional ablation lines are created by connecting the left inferior PV to the mitral annulus (mitral isthmus) and the roof of the LA between the two superior PVs. After the end of the procedure the implantable loop recorder is implanted in the parasternal area of the chest.
  Arms: Circumferential PVI
Procedure: Circumferential PVI+renal denervation — The procedure of AF ablation is the same like in the circumferential PV isolation.
  After AF ablation procedure, the angiogram of both renal arteries is performed via femoral access. After that the treatment catheter is introduced into each renal artery and is applied discrete, radiofrequency ablations lasting up to 2 min each and of 8 watts or less to obtain up to six ablations separated both longitudinally and rotationally within each renal artery. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm. After the procedure the control arterial angiogram should be done.
  Arms: Circumferential PVI+renal denervation

SUMMARY:
The purpose of this study is the comparative evaluation of systolic blood pressure (SBP) lowering, atrial fibrillation (AF) recurrence and clinical data in patients with paroxysmal/persistent AF and resistant hypertension, undergoing AF ablation alone or combined with percutaneous renal denervation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic drug-refractory AF (with history of failure of ≥2 class I or III antiarrhythmic drugs) in patients referred for catheter ablation of AF
* PAF with ≥1 monthly episodes or PersAF in patients who had already undergone ≥3 electrical cardioversions. PAF was defined as episodes lasting less than 7 days with spontaneous termination. PersAF was defined as lasting more than 7 days before being terminated pharmacologically or by electrical cardioversion.
* Office-based systolic blood pressure of ≥160 mm Hg, despite treatment with ≥3 antihypertensive drugs (including 1 diuretic)
* A glomerular filtration rate ≥45 mL/min/1⋅73 m2, with modification of diet using a renal disease formula

Exclusion Criteria:

* Previous atrial fibrillation ablation
* Type 1 of diabetes mellitus
* Structural heart disease
* Secondary cause of atrial hypertension
* Severe renal artery stenosis or renal arteries abnormalities
* Previous operations on renal arteries
* Pregnancy
* Previous heart, kidney, liver, or lung transplantation
* Unwillingness of participant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Freedom of AF or other atrial arrhythmias | 1 year

SECONDARY OUTCOMES:
Systolic blood pressure lowering | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (2):
- The Valley Health System, New York, New York, United States
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Result] Pokushalov E, Romanov A, Corbucci G, Artyomenko S, Baranova V, Turov A, Shirokova N, Karaskov A, Mittal S, Steinberg JS. A randomized comparison of pulmonary vein isolation with versus without concomitant renal artery denervation in patients with refractory symptomatic atrial fibrillation and resistant hypertension. J Am Coll Cardiol. 2012 Sep 25;60(13):1163-70. doi: 10.1016/j.jacc.2012.05.036. Epub 2012 Sep 5. PMID 22958958
- [Derived] Pokushalov E, Romanov A, Katritsis DG, Artyomenko S, Bayramova S, Losik D, Baranova V, Karaskov A, Steinberg JS. Renal denervation for improving outcomes of catheter ablation in patients with atrial fibrillation and hypertension: early experience. Heart Rhythm. 2014 Jul;11(7):1131-8. doi: 10.1016/j.hrthm.2014.03.055. Epub 2014 Mar 29. PMID 24691452